CLINICAL TRIAL: NCT04219813
Title: Urinary Gluten Detection in Patients with Non-celiac Gluten/Wheat Sensitivity
Brief Title: Urinary Gluten Immunogenic Peptides Detection in Non-celiac Gluten/Wheat Sensitivity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Pasquale Mansueto, Clinical Professor, University of Palermo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ACPM24
Record Dates: First submitted 2019-12-30; First posted 2020-01-07 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Non-celiac Gluten/Wheat Sensitivity
Keywords: Non-celiac Gluten/Wheat Sensitivity; Gluten Immunogenic Peptides; Celiac Disease
MeSH Terms: conditions — Celiac Disease | interventions — Antibody-Coated Bacteria Test, Urinary

STUDY DESIGN:
Intervention Model Description: The researchers will evaluate the urine samples of patients affected with NCGS/NCWS, diagnosed by double-blind placebo-controlled wheat challenge, on GFD. The patients will be recruited among those diagnosed in two centers: "Ambulatorio di Celiachia ed Intolleranze Alimentari" (Prof. Pasquale Mansueto) of the Geriatric Division (Director Prof. Mario Barbagallo) of the "Azienda Ospedaliera-Universitaria Paolo Giaccone'", and the "Internal Medicine Unit" (Director Prof. Antonio Carroccio) of the "Cervello-Villa Sofia" Hospital, both in Palermo, Italy. The researchers will deliver to each patient 10 kits for the analysis of the GIP and we will ask them to use them two times per week, for 5 weeks. Furthermore, the patients will test urine GIP in the event of symptoms/signs that they attribute to the accidental intake of gluten, within the same 5 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients affected with Non-celiac Gluten/Wheat Sensitivity (Other): The researchers will deliver to each patient 10 kits for the analysis of the GIP and they will ask them to use them two times per week, for 5 weeks. Furthermore, the patients will test urine GIP in the event of symptoms/signs that they attribute to the accidental intake of gluten, within the same 5 weeks. Both gastrointestinal and extra-intestinal symptoms which the patients will attribute to the accidental intake of gluten, will be considered.
  Interventions: Other: Urinary test

INTERVENTIONS:
Other: Urinary test — Detection of the presence of gluten immunogenic peptides (GIP) in the urine of NCGS/NCWS patients, evaluated two times per week, for 5 weeks, and in the event of symptoms/signs that the patients attribute to the accidental intake of gluten, within the same 5 weeks.
  Other Names: Detection of the presence of gluten immunogenic peptides (GIP) in the urine

SUMMARY:
Non-celiac gluten/wheat sensitivity (NCGS/NCWS) is a syndrome characterized by both intestinal (irritable bowel syndrome [IBS]-like presentation) and extraintestinal symptoms (headache, migraine, "foggy mind", depression, anxiety, fibromyalgia, joint and muscle pain, leg or arm numbness, eczema or skin rash), which occur after the ingestion of gluten/wheat in subjects in which celiac disease (CD) and wheat allergy diagnosis has been previously excluded. NCGS/NCWS symptoms generally occur after the ingestion of gluten/wheat, disappear within a few days of a gluten-free diet (GFD) and quickly reappear when gluten/wheat is reintroduced. A new assay, recently available on the Italian market, allows to ascertain the presence of immunogenic peptides of gluten (Gluten Immunogenic Peptides, GIP) in the urine and stool. The test might allow to ascertain if the NCGS/NCWS patients, on GFD, eat, even accidentally, gluten. Of the 2 available assays, the urinary one allows the patient himself to test the presence of GIP in relation to symptoms/signs appearing and/or social activities (e.g. meal in a restaurant). The aims of the present study are: 1) to test, in patients with NCGS/NCWS on GFD, the adherence to the elimination diet; 2) to evaluate the correlation between the symptoms' reappearance and the presence of GIP in the urine.

DETAILED DESCRIPTION:
Non-celiac gluten/wheat sensitivity (NCGS/NCWS) is a syndrome characterized by both intestinal (irritable bowel syndrome [IBS]-like presentation) and extraintestinal symptoms (headache, migraine, "foggy mind", depression, anxiety, fibromyalgia, joint and muscle pain, leg or arm numbness, eczema or skin rash), which occur after the ingestion of gluten/wheat in subjects in which celiac disease (CD) and wheat allergy diagnosis has been previously excluded. Recent data suggest that NCGS affect up to 3-6% of the general population, a higher prevalence than that reported for CD. NCGS/NCWS symptoms generally occur after the ingestion of gluten/wheat, disappear within a few days of a gluten-free diet (GFD) and quickly reappear when gluten/wheat is reintroduced. GDF is very difficult and onerous from a social (presence of gluten in many industrial food products and "contamination", both domestic and extra-domestic), psychological (e.g. for adolescents, exclusion from the "peer group", with difficulty in accepting the diagnosis) and economic point of view. A new assay, recently available on the Italian market, allows to ascertain the presence of immunogenic peptides of gluten (gluten immunogenic peptides, GIP) in the urine and stool. The test might allow to ascertain if the NCGS/NCWS patients, on GFD, eat even accidentally gluten. Of the 2 available assays, the urinary one allows the patient himself to test the presence of GIP in relation to symptoms/signs appearing and/or social activities (e.g. meal in a restaurant). The other one involves collecting a stool sample and allows to identify the gluten taken in the previous week, but it requires a laboratory, specifically equipped. To date, there are no observational studies that indicate the performance of the test in patients with NCGS/NCWS. The aims of the present study are: 1) to test, in patients with NCGS/NCWS on GFD, the adherence to the elimination diet; 2) to evaluate the correlation between the symptoms' reappearance and the presence of GIP in the urine.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from NCGS/NCWS on Gluten-Free Diet (GFD).

Exclusion Criteria:

* celiac patients or those suffering from IgE-mediated gluten/wheat allergy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to GFD of NCGS/NCWS patients | 24 months
  The researchers will evaluate the adherence to Gluten-Free Diet (GFD) of NCGS/NCWS patients on GFD by the absence/presence of gluten immunogenic peptides (GIP) in their urine samples.

SECONDARY OUTCOMES:
Gastrointestinal and extraintestinal symptoms/signs reappearance | 24 months
  The researchers will evaluate the correlation between gastrointestinal (evaluated by the Gastrointestinal Symptom Rating Scale, GSRS) and/or extraintestinal (evaluated by an ad hoc Scale) symptoms/signs reappearance and the presence of gluten immunogenic peptides (GIP) in the urine of NCGS/NCWS patients on Gluten-Free Diet (GFD), by possible accidental intake.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carroccio, PHD, Principal Investigator — University of Palermo
Locations (2):
- Italy (2):
  - Department of Internal Medicine, University Hospital of Palermo, Palermo, Palermo
  - Internal Medicine Division of the "Cervello-Villa Sofia" Hospital, Palermo, PA

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carroccio A, D'Alcamo A, Cavataio F, Soresi M, Seidita A, Sciume C, Geraci G, Iacono G, Mansueto P. High Proportions of People With Nonceliac Wheat Sensitivity Have Autoimmune Disease or Antinuclear Antibodies. Gastroenterology. 2015 Sep;149(3):596-603.e1. doi: 10.1053/j.gastro.2015.05.040. Epub 2015 May 27. PMID 26026392
- [Background] Carroccio A, Mansueto P, D'Alcamo A, Iacono G. Non-celiac wheat sensitivity as an allergic condition: personal experience and narrative review. Am J Gastroenterol. 2013 Dec;108(12):1845-52; quiz 1853. doi: 10.1038/ajg.2013.353. Epub 2013 Nov 5. PMID 24169272
- [Background] Carroccio A, Mansueto P, Iacono G, Soresi M, D'Alcamo A, Cavataio F, Brusca I, Florena AM, Ambrosiano G, Seidita A, Pirrone G, Rini GB. Non-celiac wheat sensitivity diagnosed by double-blind placebo-controlled challenge: exploring a new clinical entity. Am J Gastroenterol. 2012 Dec;107(12):1898-906; quiz 1907. doi: 10.1038/ajg.2012.236. Epub 2012 Jul 24. PMID 22825366
- [Background] Carroccio A, Rini G, Mansueto P. Non-celiac wheat sensitivity is a more appropriate label than non-celiac gluten sensitivity. Gastroenterology. 2014 Jan;146(1):320-1. doi: 10.1053/j.gastro.2013.08.061. Epub 2013 Nov 22. No abstract available. PMID 24275240
- [Background] Catassi C, Elli L, Bonaz B, Bouma G, Carroccio A, Castillejo G, Cellier C, Cristofori F, de Magistris L, Dolinsek J, Dieterich W, Francavilla R, Hadjivassiliou M, Holtmeier W, Korner U, Leffler DA, Lundin KE, Mazzarella G, Mulder CJ, Pellegrini N, Rostami K, Sanders D, Skodje GI, Schuppan D, Ullrich R, Volta U, Williams M, Zevallos VF, Zopf Y, Fasano A. Diagnosis of Non-Celiac Gluten Sensitivity (NCGS): The Salerno Experts' Criteria. Nutrients. 2015 Jun 18;7(6):4966-77. doi: 10.3390/nu7064966. PMID 26096570
- [Background] Di Liberto D, Mansueto P, D'Alcamo A, Lo Pizzo M, Lo Presti E, Geraci G, Fayer F, Guggino G, Iacono G, Dieli F, Carroccio A. Predominance of Type 1 Innate Lymphoid Cells in the Rectal Mucosa of Patients With Non-Celiac Wheat Sensitivity: Reversal After a Wheat-Free Diet. Clin Transl Gastroenterol. 2016 Jul 7;7(7):e178. doi: 10.1038/ctg.2016.35. PMID 27388423
- [Background] Drossman DA. Functional Gastrointestinal Disorders: History, Pathophysiology, Clinical Features and Rome IV. Gastroenterology. 2016 Feb 19:S0016-5085(16)00223-7. doi: 10.1053/j.gastro.2016.02.032. Online ahead of print. PMID 27144617
- [Background] Losurdo G, Principi M, Iannone A, Giangaspero A, Piscitelli D, Ierardi E, Di Leo A, Barone M. Predictivity of Autoimmune Stigmata for Gluten Sensitivity in Subjects with Microscopic Enteritis: A Retrospective Study. Nutrients. 2018 Dec 18;10(12):2001. doi: 10.3390/nu10122001. PMID 30567296
- [Background] Mansueto P, Seidita A, D'Alcamo A, Carroccio A. Non-celiac gluten sensitivity: literature review. J Am Coll Nutr. 2014;33(1):39-54. doi: 10.1080/07315724.2014.869996. PMID 24533607
- [Background] Sapone A, Bai JC, Ciacci C, Dolinsek J, Green PH, Hadjivassiliou M, Kaukinen K, Rostami K, Sanders DS, Schumann M, Ullrich R, Villalta D, Volta U, Catassi C, Fasano A. Spectrum of gluten-related disorders: consensus on new nomenclature and classification. BMC Med. 2012 Feb 7;10:13. doi: 10.1186/1741-7015-10-13. PMID 22313950